CLINICAL TRIAL: NCT04741750
Title: Does a Simplified Algorithm and Integrated HCV Care Improve Linkage to Care, Retention, and Cure Among People Who Inject Drugs? A Pragmatic Quality Improvement Randomized Controlled Trial
Brief Title: Increasing HCV Linkage to Care Among People Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Family Health Centers of San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GSHCV
Record Dates: First submitted 2021-01-19; First posted 2021-02-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Hepatitis C treatment; People who inject drugs; Mobile medical clinic; People experiencing homelessness; Treatment initiation; Linkage to care; Quality improvement
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: A pragmatic quality improvement randomized controlled trial will be conducted among 200 people who inject drugs (PWID) with chronic hepatitis C virus (HCV), age ≥18 years, recruited from Family Health Centers of San Diego's mobile clean syringe exchange program (CSEP). Patients will be recruited to undergo HCV testing. Patients with a positive HCV Ab rapid finger stick test will be randomly allocated (ratio 1:1) to receiving treatment immediately in a mobile medical clinic (n=100) or in a community clinic (n=100, this will serve as a concurrent control group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation is concealed until intervention is assigned. The PI and those analyzing the outcome of the trial will remain blinded throughout the entirety of the study. Only the patients and those delivering the intervention will be aware of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care within Community Clinics (No Intervention): Complete blood count, comprehensive metabolic panel, international normalized ratio, HCV RNA, hepatitis B virus (HBV) serologies, point of care HIV test, and point of care liver fibrosis measurement. HCV genotype if required by patient's insurance for prior authorization. Care for opioid use disorder and skin infection is offered. Completion of the initial visit workup is sufficient to initiate a prior authorization request for DAAs from payers and an appointment for MAT follow-up in a community clinic if indicated. Patient coordination; authorization with insurance companies; scheduling appointments, follow-up, and ancillary support services will be conducted by a Patient Navigator. Patients are seen every 2-4 weeks for monitoring and adherence support. HCV treatment regimens are at the discretion of the treating provider in accordance with AASLD/IDSA guidelines and insurance requirements. Twelve weeks after HCV therapy completion, SVR12 HCV RNA and SVR12 CMP tests will be obtained.
- Simplified Care within a Mobile Medical Unit (Experimental): Simplified Care treatment is the same as for Usual Care with the exception that it is taking place within a mobile medical clinic that is scheduled to deliver treatment in alignment with regular syringe exchange services.
  Interventions: Other: Simplified HCV care within a mobile medical unit

INTERVENTIONS:
Other: Simplified HCV care within a mobile medical unit — Delivers guideline-based care for HCV in a stream-lined manner on a mobile medical unit
  Arms: Simplified Care within a Mobile Medical Unit

SUMMARY:
Our study will test the effectiveness of a simplified approach to delivering Hepatitis C Virus (HCV) care in a street-based mobile medical clinic among people who inject drugs in increasing treatment initiation, retention, and cure. Rates of HCV treatment initiation, retention, and cure will be compared between patients offered the simplified approach to delivering HCV care in a mobile medical clinic versus those who are linked to a community clinic delivering a current practice of usual care. The investigators hypothesize that the simplified approach to delivering HCV care in a street-based mobile medical clinic will result in higher treatment initiation, retention, and cure than the current practice of usual care in community clinics.

DETAILED DESCRIPTION:
With as many as 2.4 million Americans affected by chronic Hepatitis C Virus (HCV), it is one of the most common blood-borne diseases in the United States. Nationwide, rates of new infections have risen dramatically among young adults in their 20s and 30s, the same cohorts most affected by the opioid epidemic, with as many as 70% of new infections related to injection drug use. Local/regional rates of new infection mirror these national surveillance findings. In San Diego, between 2011 and 2016, women aged 20-29 experienced a 62.2% increase in new HCV infections, while new infections among men aged 20-29 spiked 46.6%, with injection drug use cited as the most common form of transmission. Expanded prevalence estimates indicate a population prevalence rate for HCV of 2.0% to 2.7% in San Diego County, suggesting that approximately 65,000 to 88,000 individuals in the region are likely HCV-infected. These alarming increases in new HCV infections demand effective treatment delivered to populations that historically have been difficult to reach and are characterized by disparities in HCV screening, linkage to care, and treatment access due to a constellation of barriers to care. Advances in HCV treatment and care (e.g., the development of highly effective direct-acting antivirals--DAAs) show promise for treating these populations and have led to worldwide HCV elimination goals, as well as local/regional elimination campaigns. While the American Association for the Study of Liver Diseases/Infectious Diseases Society of America (AASLD/IDSA)'s guidelines have long been considered the gold standard for HCV diagnosis, workup, and treatment (and remain appropriate for HCV specialists, especially in complex cases of HCV infection) recent World Health Organization (WHO) HCV guidelines and published consensus statements call for implementation of streamlined and simplified algorithms for HCV care, delivered in an integrated primary care setting. They highlight that most patients, particularly younger people who inject drugs (PWID), have a low risk of cirrhosis, do not require genotyping if treated with pangenotypic regimens, and may be lost to follow-up due to overly complex, time-intensive, and costly evaluations. Furthermore, emerging evidence indicates that PWID achieve the same high cure rates as non-injection drug user patients when treated with DAAs. While research indicates that DAAs have high efficacy and safety and can now be used by primary care providers to treat HCV there are still groups, especially PWID, who experience treatment disparities due to access and treatment barriers. Limited evidence exists to support the effectiveness of expanding screening and treatment access via the use of mobile medical clinics co-located with services for PWID. Only one study to date has shown that point of care testing in a mobile medical clinic resulted in significantly higher rates of HCV infected patients being linked to HCV treatment in 30 days compared to standard phlebotomy HCV testing. Therefore, the proposed study will test the effectiveness of a simplified HCV algorithm with integrated care (including the offer of buprenorphine prescriptions and abscess care), in a street-based mobile clinic setting among PWID, in increasing treatment initiation and retention rates. Rates of HCV treatment initiation and retention will be compared between patients offered a simplified HCV care in a mobile medical clinic versus those who are linked to the current practice of usual care in community clinics.

ELIGIBILITY:
Inclusion Criteria: Participants will be positive HCV antibody and positive HCV RNA patients aged 18 years or older who are willing to undergo HCV treatment.

Exclusion Criteria: There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who initiate HCV treatment | 6 months of follow-up
  Initiating treatment with a Direct-Acting Antiviral (DAA)

SECONDARY OUTCOMES:
Number of patients who complete HCV treatment | 16 weeks after treatment initiation
  Completing a full treatment course of 8 or 12 weeks of DAA therapy
SVR12 rates | At least 12 weeks following DAA completion
  Undetectable HCV RNA on or after the SVR12 time point
Initiation rates for medication-assisted treatment (MAT) for Opioid Use Disorder | During the first 3 months of follow-up after enrollment
  Attendance of at least one visit to a community clinic for treatment of Opioid Use Disorder
Persistent rate for MAT | During 6 months of follow-up after enrollment
  > 3 visits for MAT
Number of patients who receive abscess care | During 6 months of follow-up after enrollment
  Treatment for skin infection or abscess
Prevalence of engagement in care | During 6 months of follow-up after enrollment
  The number of visits for any reason during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Family Health Centers of San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramers CB, Vawter N, Northrup A, Klaman SL, Lewis SV, Tam A, Del Aguila C, Lewis R, Mendez B, Reyes L, Matthews E, Rojas S, Godino JG. Simplified and Integrated Hepatitis C Virus Testing and Treatment Algorithm for Unhoused People Who Inject Drugs. Open Forum Infect Dis. 2025 May 22;12(6):ofaf302. doi: 10.1093/ofid/ofaf302. eCollection 2025 Jun. PMID 40476033
- [Derived] Klaman SL, Godino JG, Northrup A, Lewis SV, Tam A, Carrillo C, Lewis R, Matthews E, Mendez B, Reyes L, Rojas S, Ramers C. Does a simplified algorithm and integrated HCV care model improve linkage to care, retention, and cure among people who inject drugs? A pragmatic quality improvement randomized controlled trial protocol. BMC Infect Dis. 2024 Jan 19;24(1):105. doi: 10.1186/s12879-024-08982-1. PMID 38238686